CLINICAL TRIAL: NCT04022603
Title: Impact of High-level Oxygen Therapy on the Reconditioning of Type I Hypoxemic Respiratory Insufficiency Patients in Intensive Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr David DE BELS (Other)
Responsible Party: Sponsor-Investigator, Dr David DE BELS, Head of intensive care unit, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUB-BPCO
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Hypoxemic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optiflow nasal googles (Experimental): Oxygen provided by means of high throughput nasal googles (Optiflow, Fisher&Paykel- New Zealand).
  Interventions: Device: Cyclometer Ergometer
- Venturi mask (Active Comparator): Oxygen provided by means of a Venturi mask.
  Interventions: Device: Cyclometer Ergometer

INTERVENTIONS:
Device: Cyclometer Ergometer — The measurements are carried out on a max effort of 12 minutes on a cyclometer ergometer with a constant load (Motomed viva2 light). A first effort is made with a Venturi type mask whose Inspired Fraction in Oxygen (FiO2) is set for a pulsated oxygen saturation (SpO2) greater than or equal to 85%, and then a second at 2h interval with high-throughput googles (Optiflow) with the corresponding FiO2.

SUMMARY:
High-throughput oxygen therapy is known as an alternative to non-invasive ventilation, with a benefit in terms of survival in non-hypercapnic respiratory failure patients.

The use of high-throughput oxygen therapy is well studied in stable chronic obstructive pulmonary disease (COPD) patients and has as known effects the decrease of transcutaneous CO2 and respiratory rate, and the increase in the inspiratory/expiratory time report, in the tidal volume and in the forced expiratory volume per second.

In the event of an exacerbation, high-flow oxygen therapy has shown to be beneficial in terms of increased mean airway pressure, tidal volume with a decrease in hypercapnia, and respiratory rate.

The net effect on the CO2 pressure is linked to the CO2 clearance of the dead anatomical space by the high throughput. The effect can be compared with the one of non invasive ventilation in a stable COPD patient.

Oxygen therapy, even in patients with non-hypoxic COPD at rest, has benefits in terms of performance and improvement of quality of life. High-throughput oxygen therapy has also shown a benefit in COPD patients in revalidation units, in terms of exercise performance and oxygenation.

However, the reconditioning of critical patients in acute situations, by means of nasal goggles, has never been studied.

ELIGIBILITY:
Inclusion Criteria:

* Acute respiratory insufficiency type I, oxygen partial pressure (PaO2) <60 mmHg under oxygen without hypercapnia.
* Invasive arterial pressure measure

Exclusion Criteria:

* Hemodynamic instability
* Patient under continuous high throughput oxygen therapy
* Left cardiac insufficiency
* Arteritis of the lower limbs
* Neuromuscular pathology
* Osteo-articular limitations
* Hemoglobin inferior to 8g/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-08-03 (Actual)

PRIMARY OUTCOMES:
Pulsated oxygen saturation (Sp02) | Baseline
  SpO2 is an estimate of the amount of oxygen in the blood. More precisely, it represents the percentage of oxygenated hemoglobin (containing oxygen) relative to the total amount of hemoglobin in the blood (oxygenated hemoglobin and non-oxygenated hemoglobin).
Pulsated oxygen saturation (Sp02) | 12 minutes (maximal effort)
  SpO2 is an estimate of the amount of oxygen in the blood. More precisely, it represents the percentage of oxygenated hemoglobin (containing oxygen) relative to the total amount of hemoglobin in the blood (oxygenated hemoglobin and non-oxygenated hemoglobin).
Oxygen inspired fraction (FiO2) | Baseline
  Oxygen inspired fraction (FiO2) is the fraction or percentage of oxygen present in the gas mixture that a person breathes.
Oxygen inspired fraction (FiO2) | 12 minutes (maximal effort)
  Oxygen inspired fraction (FiO2) is the fraction or percentage of oxygen present in the gas mixture that a person breathes.
Blood gasometry | Baseline
  Arterial blood analysis
Blood gasometry | 12 minutes (maximal effort)
  Arterial blood analysis
Heart rate | Baseline
  The heart rate is the number of heartbeats per unit minute.
Heart rate | 12 minutes (maximal effort)
  The heart rate is the number of heartbeats per minute.
Respiratory rate | Baseline
  Number of breath cycles (inspiration and expiration) per minute.
Respiratory rate | 12 minutes (maximal effort)
  Number of breath cycles (inspiration and expiration) per minute.
Mean arterial pressure | Baseline
  Mean arterial pressure
Mean arterial pressure | 12 minutes (maximal effort)
  Mean arterial pressure
Systolic blood pressure | Baseline
  Systolic blood pressure (pressure in the artery as the heart contracts)
Systolic blood pressure | 12 minutes (maximal effort)
  Systolic blood pressure (pressure in the artery as the heart contracts)
Borg score | 12 minutes (maximal effort)
  The Borg scale is a quantitative measure of the perception of effort during exercise. The scale between 0 and 10 was designed to approximate the heart rate of a healthy young adult (effort 8 represents 80% of the cardiac frequency).
Forced expiratory volume per second (FEV1) | Baseline
  The "Forced Expiratory Volume Per Second" (FEV1) is the volume of air exhaled during the first second of a so-called "forced" exhalation, following deep inspiration. It is measured by spirometry.
Functional residual capacity (CFR) | Baseline
  Volume of air remaining in the airways after a spontaneous expiration (not forced)

SECONDARY OUTCOMES:
Age | Baseline
  Age
Weight | Baseline
  Weight
Sex | Baseline
  Sex

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Redant, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No